CLINICAL TRIAL: NCT01686750
Title: A Cluster Randomized Trial of Integrated Care Centers to Improve Access to HIV Prevention, Testing, and Treatment Services Among High-Risk Vulnerable Populations in India
Brief Title: Integrated Care Centers to Improve HIV Outcomes in Vulnerable Indian Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); YR Gaitonde Centre for AIDS Research and Education (Other); Elton John AIDS Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00047702; R01DA032059 (NIH); R01MH089266 (NIH)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: HIV Infection
Keywords: HIV; injection drug use; men who have sex with men; voluntary counselling and testing; risk reduction; sexually transmitted infections; community viral load; antiretroviral therapy
MeSH Terms: conditions — HIV Infections; Homosexuality; Risk Reduction Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated care centers (Experimental): Integrated care centers will provide HIV prevention and treatment services to high risk populations of IDU or MSM in an accepting and supportive environment.
  * HIV voluntary counseling and testing & staging
  * Risk reduction services including free condoms, needle and syringe exchange, opiate substitution therapy
  * Substance abuse counseling
  * Sexually transmitted infection screening and treatment
  * Access to free antiretroviral therapy and adherence support
  * Peer community outreach
  Interventions: Behavioral: Integrated care centers
- Standard services (No Intervention): In Standard Services sites, HIV testing, prevention, and treatment services will be available through standard venues. Government centers typically provide most HIV testing services and are the only source for free antiretroviral therapy. Non-governmental organizations typically provide prevention and risk reduction services.

INTERVENTIONS:
Behavioral: Integrated care centers
  Arms: Integrated care centers

SUMMARY:
This is a cluster randomized trial to evaluate the effectiveness of integrated care centers (ICC) to improve access to HIV testing, prevention services, and treatment among high-risk populations of injection drug users (IDU) and men who have sex with men (MSM) in India. We will collect baseline ethnographic and survey data from approximately 27 IDU or MSM sites in India. We will use baseline data to select 22 sites for the trial (12 IDU and 10 MSM) and to stratify sites according to key baseline characteristics. We will perform stratified randomization to assign sites to either the ICC intervention or to standard services. ICCs, which will be either IDU or MSM-focused, will provide an accepting atmosphere in which members of vulnerable groups can drop-in, receive rapid HIV voluntary counselling and testing, risk reduction counseling and services, and antiretroviral therapy. ICCs will be scaled-up from existing governmental or non-governmental organizations and services provided at ICCs will be supported by the National AIDS Control Organization (NACO) of India. After providing services in communities for two years, we will conduct an evaluation survey (with biological and behavioral measures) of approximately 1000 subjects in the target populations in each of the 22 study sites. Integrated care centers have the potential to improve access to HIV prevention and treatment services among vulnerable, high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

Key Informant Interviews:

Persons may be included in the key informant interviews if they meet all of the following criteria:

1. 18 years of age or older
2. Knowledge of the local HIV risk group of interest (IDU or MSM)
3. Psychologically fit to participate in the study and to understand the consent
4. Ability to comprehend one of the consent translation languages
5. Provide informed consent

Focus groups:

Persons may be included in the focus groups if they meet all of the following criteria:

1. 18 years of age or older
2. Member of a target HIV risk group, meeting criterion 2a or 2b

   1. IDU: self-reported injection drug use in prior 12 months
   2. MSM: self-identify as male and report oral/anal sex with another male in prior 12 months
3. Psychologically fit to participate in the study and to understand the consent
4. Ability to comprehend one of the consent translation languages
5. Provide informed consent

Baseline or evaluation respondent-driven sampling (RDS) survey

Persons may be included in the baseline or evaluation RDS survey if they meet all of the following criteria:

1. 18 years of age or older
2. Member of a target HIV risk group, meeting criterion 2a or 2b

   1. IDU: self-reported injection drug use in prior 24 months
   2. MSM: self-identify as male and report oral/anal sex with another male in prior 12 months
3. Psychologically fit to participate in the study and to understand the consent
4. Ability to comprehend one of the consent translation languages
5. Present a valid RDS referral coupon (unless a seed)
6. Provide informed consent

Exclusion Criteria:

Key Informant Interviews:

Persons will be excluded from the key informant interviews if they meet any of the following criteria:

1. Younger than 18 years
2. Do not have knowledge of the local HIV risk group of interest (IDU or MSM)
3. Are not psychologically fit to participate in the study or to understand the consent
4. Do not have ability to comprehend one of the consent translation languages
5. Do not provide informed consent

Focus groups:

Persons will be excluded from the focus groups if they meet any of the following criteria:

1. Younger than 18 years
2. Are not a member of a target HIV risk group, meeting neither criterion 2a nor 2b

   1. IDU: self-reported injection drug use in prior 12 months
   2. MSM: self-identify as male and report oral/anal sex with another male in prior 12 months
3. Are not psychologically fit to participate in the study or to understand the consent
4. Do not have ability to comprehend one of the consent translation languages
5. Do not provide informed consent

Baseline or evaluation RDS survey

Persons will be excluded in the baseline or evaluation RDS survey if they meet any of the following criteria:

1. Younger than 18 years
2. Are not a member of a target HIV risk group, meeting neither criterion 2a nor 2b

   1. IDU: self-reported injection drug use in prior 24 months
   2. MSM: self-identify as male and report oral/anal sex with another male in prior 12 months
3. Are not psychologically fit to participate in the study or to understand the consent
4. Do not have ability to comprehend one of the consent translation languages
5. Do not present a valid RDS referral coupon and are not a seed
6. Do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21726 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Lucas, MD, Principal Investigator — Johns Hopkins University; Shruti Mehta, PhD, Principal Investigator — Johns Hopkins University; David D Celentano, ScD, Principal Investigator — Johns Hopkins University; Suniti Solomon, MD, Principal Investigator — YR Gaitonde Centre for AIDS Research and Education; Aylur Srikrishnan, BA, Principal Investigator — YR Gaitonde Centre for AIDS Research and Education; Suresh Kumar, MPH, Principal Investigator — YR Gaitonde Centre for AIDS Research and Education; Sunil S Solomon, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- YR Gaitonde Center for AIDS Research and Education, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Solomon SS, Mehta SH, Srikrishnan AK, Vasudevan CK, Mcfall AM, Balakrishnan P, Anand S, Nandagopal P, Ogburn EL, Laeyendecker O, Lucas GM, Solomon S, Celentano DD. High HIV prevalence and incidence among MSM across 12 cities in India. AIDS. 2015 Mar 27;29(6):723-31. doi: 10.1097/QAD.0000000000000602. PMID 25849835
- [Background] Lucas GM, Solomon SS, Srikrishnan AK, Agrawal A, Iqbal S, Laeyendecker O, McFall AM, Kumar MS, Ogburn EL, Celentano DD, Solomon S, Mehta SH. High HIV burden among people who inject drugs in 15 Indian cities. AIDS. 2015 Mar 13;29(5):619-28. doi: 10.1097/QAD.0000000000000592. PMID 25715105
- [Background] Solomon SS, Mehta SH, Srikrishnan AK, Solomon S, McFall AM, Laeyendecker O, Celentano DD, Iqbal SH, Anand S, Vasudevan CK, Saravanan S, Lucas GM, Kumar MS, Sulkowski MS, Quinn TC. Burden of hepatitis C virus disease and access to hepatitis C virus services in people who inject drugs in India: a cross-sectional study. Lancet Infect Dis. 2015 Jan;15(1):36-45. doi: 10.1016/S1473-3099(14)71045-X. Epub 2014 Dec 3. PMID 25486851
- [Background] Solomon SS, Lucas GM, Celentano DD, Sifakis F, Mehta SH. Beyond surveillance: a role for respondent-driven sampling in implementation science. Am J Epidemiol. 2013 Jul 15;178(2):260-7. doi: 10.1093/aje/kws432. Epub 2013 Jun 25. PMID 23801014
- [Background] Solomon SS, Lucas GM, Celentano DD, McFall AM, Ogburn E, Moulton LH, Srikrishnan AK, Kumar MS, Anand S, Solomon S, Mehta SH. Design of the Indian NCA study (Indian national collaboration on AIDS): a cluster randomized trial to evaluate the effectiveness of integrated care centers to improve HIV outcomes among men who have sex with men and persons who inject drugs in India. BMC Health Serv Res. 2016 Nov 14;16(1):652. doi: 10.1186/s12913-016-1905-5. PMID 27842543
- [Background] Mehta SH, Lucas GM, Solomon S, Srikrishnan AK, McFall AM, Dhingra N, Nandagopal P, Kumar MS, Celentano DD, Solomon SS. HIV care continuum among men who have sex with men and persons who inject drugs in India: barriers to successful engagement. Clin Infect Dis. 2015 Dec 1;61(11):1732-41. doi: 10.1093/cid/civ669. Epub 2015 Aug 6. PMID 26251048
- [Result] Solomon SS, Solomon S, McFall AM, Srikrishnan AK, Anand S, Verma V, Vasudevan CK, Balakrishnan P, Ogburn EL, Moulton LH, Kumar MS, Sachdeva KS, Laeyendecker O, Celentano DD, Lucas GM, Mehta SH; Indian National Collaboration on AIDS Study. Integrated HIV testing, prevention, and treatment intervention for key populations in India: a cluster-randomised trial. Lancet HIV. 2019 May;6(5):e283-e296. doi: 10.1016/S2352-3018(19)30034-7. Epub 2019 Apr 2. PMID 30952565
- [Derived] Prabhu S, Mehta SH, McFall AM, Srikrishnan AK, Vasudevan CK, Lucas GM, Celentano DD, Solomon SS. Substance use is associated with condomless anal intercourse among men who have sex with men in India: a partner-level analysis. BMC Public Health. 2022 Apr 11;22(1):722. doi: 10.1186/s12889-022-13192-y. PMID 35410326
- [Derived] Solomon SS, Quinn TC, Solomon S, McFall AM, Srikrishnan AK, Verma V, Kumar MS, Laeyendecker O, Celentano DD, Iqbal SH, Anand S, Vasudevan CK, Saravanan S, Thomas DL, Sachdeva KS, Lucas GM, Mehta SH. Integrating HCV testing with HIV programs improves hepatitis C outcomes in people who inject drugs: A cluster-randomized trial. J Hepatol. 2020 Jan;72(1):67-74. doi: 10.1016/j.jhep.2019.09.022. Epub 2019 Oct 8. PMID 31604081
- [Derived] Solomon SS, Mehta SH, McFall AM, Srikrishnan AK, Saravanan S, Laeyendecker O, Balakrishnan P, Celentano DD, Solomon S, Lucas GM. Community viral load, antiretroviral therapy coverage, and HIV incidence in India: a cross-sectional, comparative study. Lancet HIV. 2016 Apr;3(4):e183-90. doi: 10.1016/S2352-3018(16)00019-9. Epub 2016 Mar 11. PMID 27036994

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited by respondent-driven sampling in 22 sites in India.
Units Other Than Participants: Clusters
Groups:
- Integrated Care Centers: Integrated care centers will provide HIV prevention and treatment services to high risk populations of injecting drug users (IDU) or MSM in an accepting and supportive environment.
  * HIV voluntary counseling and testing & staging
  * Risk reduction services including free condoms, needle and syringe exchange, opiate substitution therapy
  * Substance abuse counseling
  * Sexually transmitted infection screening and treatment
  * Access to free antiretroviral therapy and adherence support
  * Peer community outreach
Period: Overall Study
Arm/Group | Integrated Care Centers | Standard Services
Started | 11001; 11 Clusters | 10725; 11 Clusters
Completed | 11001; 11 Clusters | 10725; 11 Clusters
Not Completed | 0; 0 Clusters | 0; 0 Clusters

BASELINE CHARACTERISTICS:
Units Other Than Participants: Clusters
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care Centers | Standard Services | Total
Number analyzed (Participants) | 11001 | 10725 | 21726
Number analyzed (Clusters) | 11 | 11 | 22
Age, Continuous [Median (Full Range); unit: years] | 30 [24 to 34] | 29 [26 to 35] | 29 [24 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 272 | 493
  Male | 10780 | 10453 | 21233
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11001 | 10725 | 21726
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
At least secondary school education [Count of Participants; unit: Participants] — Participants who have had at least a secondary school education.
  Participants | 8729 | 7455 | 16184

OUTCOME MEASURES:

1. Primary Outcome: Proportion Reporting HIV Testing in the Prior 12 Months
Description: Self-reported HIV testing in the prior 12 months among all survey participants, excluding those who reported being diagnosed with HIV more than 12 months previously.
Time Frame: 2 years
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 11001 | 10725
Number analyzed (clusters) | 11 | 11
percentage of participants | 36.9 [20.5 to 53.3] | 26.2 [4.7 to 37.3]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; We compared the sampling-weighted prevalence of outcomes at Integrated Care Centers (ICCs) and usual care from the evaluation survey. We used linear regression models that had terms for intervention status (integrated care vs usual care), stratum (PWID and MSM), and the baseline proportion of the outcome being assessed. Site-level proportions from both evaluation and baseline respondent-driven sampling were log transformed before being entered into the regression model; Test type: Superiority; p = 0.09, Prevalence ratio; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.95 to 1.81] — Therefore, the exponentiated coefficients for intervention status represent the prevalence ratio with 95% confidence interval (CI) and are interpreted as the relative percentage difference in the outcome associated with the intervention

2. Secondary Outcome: Proportion of HIV-infected Participants Aware of Status
Description: Proportion of HIV-positive participants that were aware of their status at the time of the visit
Time Frame: 2 years
Population: Participants who tested HIV-positive at the survey visit
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 1974 | 2306
Number analyzed (clusters) | 11 | 11
percentage of participants | 65.2 [24 to 86.5] | 59.4 [14.4 to 97.4]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.80 to 1.50]

3. Secondary Outcome: Proportion of HIV-infected Participants Visiting an HIV Treatment Provider in Prior 6 Months
Time Frame: 2 years
Population: HIV-positive survey participants
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Groups:
- Integrated Care Centers: Integrated care centers will provide HIV prevention and treatment services to high risk populations of IDU or MSM in an accepting and supportive environment.
  * HIV voluntary counseling and testing & staging
  * Risk reduction services including free condoms, needle and syringe exchange, opiate substitution therapy
  * Substance abuse counseling
  * Sexually transmitted infection screening and treatment
  * Access to free antiretroviral therapy and adherence support
  * Peer community outreach
  Integrated care centers
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 1974 | 2306
Number analyzed (clusters) | 11 | 11
percentage of participants | 45.7 [3.5 to 73.9] | 40.8 [3.1 to 88.0]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.61 to 1.81]

4. Secondary Outcome: Proportion of Antiretroviral Therapy-eligible HIV-infected Participants Using Antiretroviral Therapy
Time Frame: 2 years
Population: HIV-positive participants that meet criteria for antiretroviral therapy in India at the time of the study
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 1647 | 1749
Number analyzed (clusters) | 11 | 11
percentage of participants | 57 [11.4 to 87] | 46.8 [2 to 95.1]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.77 to 2.41]

5. Secondary Outcome: Community Viral Load
Description: Average log(10) HIV RNA concentration among HIV-infected participants
Time Frame: 2 years
Population: Samples were not collected therefore there is no data to report.
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion of HIV-infected Participants With Suppressed HIV RNA
Description: Proportion of HIV-positive participants meeting criteria for antiretroviral therapy [cluster of differentiation 4 (CD4) count <350 cells/mm3 or current or past use of antiretroviral therapy)] who have a suppressed viral load (HIV RNA <150 copies/mL)
Time Frame: 2 years
Population: HIV-positive participants who meet criteria for antiretroviral therapy
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 1647 | 1749
Number analyzed (clusters) | 11 | 11
percentage of participants | 47.3 [6.7 to 78.6] | 46.7 [7.4 to 82.9]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.65 to 1.28]

7. Secondary Outcome: Prevalence of Recent HIV Infection
Time Frame: 2 years
Population: Samples were not collected therefore there is no data to report.
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Proportion of IDU Reporting Needle or Syringe Sharing in Prior 6 Months
Time Frame: 2 years
Population: Participants from the PWID sites
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 6000 | 5721
Number analyzed (clusters) | 6 | 6
percentage of participants | 30.1 [2.4 to 30.8] | 31.8 [6.8 to 56.9]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio, log = 1.44, 95% CI 2-sided [0.42 to 4.93]

9. Secondary Outcome: Proportion of IDU Reporting Drug Abstinence in Prior 6 Months
Time Frame: 2 years
Population: Participants at PWID sites
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 6000 | 5721
Number analyzed (clusters) | 6 | 6
percentage of participants | 28.2 [10.4 to 72.9] | 16.5 [1.7 to 42.3]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio, log = 1.87, 95% CI 2-sided [0.49 to 7.16]

10. Secondary Outcome: Proportion of MSM Reporting Unprotected Anal Intercourse With Non-main Partner in Prior 6 Months
Time Frame: 2 years
Population: Participants at MSM sites
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 5001 | 5004
Number analyzed (clusters) | 5 | 5
percentage of participants | 56.2 [39.8 to 78.9] | 69.3 [41.7 to 84]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.53 to 1.56]

11. Secondary Outcome: Number of Non-main Male Partners in Prior 6 Months in MSM
Time Frame: 2 years
Population: Participants at MSM sites
Measure: Mean (Full Range); unit: partners
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 5001 | 5004
Number analyzed (clusters) | 5 | 5
partners | 3.0 [0.6 to 6.4] | 3.1 [1.5 to 8.0]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-4.2 to 4.2]

12. Secondary Outcome: Proportion Reporting Substance Abuse Among MSM
Time Frame: 2 years
Population: Samples were not collected therefore there is no data to report.
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Proportion With Depressive Symptoms
Description: Participants with Score >=10 on Patient Health Questionnaire-9
Time Frame: 2 years
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 11001 | 10725
Number analyzed (clusters) | 11 | 11
percentage of participants | 13.4 [1.2 to 26.9] | 18.2 [3.7 to 35.1]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.47 to 1.52]

14. Secondary Outcome: Number of Unprotected Sexual Acts Reported by MSM
Time Frame: 2 years
Population: Samples were not collected therefore there is no data to report.
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Vicarious Stigma as Assessed by 6-item Stigma Scale
Description: Summed score from a 6-item stigma scale (range 0-18), with higher values indicating more perceived stigma
Time Frame: 2 years
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 11001 | 10725
Number analyzed (clusters) | 11 | 11
score on a scale | 2.9 [2.1 to 4.2] | 4.6 [1.5 to 7.1]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.0 to -0.6]

16. Secondary Outcome: Proportion Reporting Spouse Ever Tested for HIV
Time Frame: 2 years
Population: Participants with a spouse (opposite sex)
Measure: Mean (Full Range); unit: percentage of participants
Units Other Than Participants: clusters
Arm/Group | Integrated Care Centers | Standard Services
Number analyzed (Participants) | 5550 | 4439
Number analyzed (clusters) | 11 | 11
percentage of participants | 45.9 [19.2 to 74.3] | 46.8 [7.7 to 79.9]
Statistical Analysis 1: Comparison: Integrated Care Centers vs Standard Services; Test type: Superiority; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.64 to 1.36]

ADVERSE EVENTS:
Time Frame: This study was based on cross-sectional surveys. Therefore adverse events were only documented at the time of the survey visit (1 day).
Arm/Group | Integrated Care Centers | Standard Services
All-Cause Mortality (participants affected / at risk) | 0/11001 | 0/10725
Serious Adverse Events (participants affected / at risk) | 0/11001 | 0/10725
Other Adverse Events (participants affected / at risk) | 0/11001 | 0/10725

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT01686750/Prot_SAP_000.pdf